CLINICAL TRIAL: NCT05113251
Title: A Phase 3 Open-label Trial of Neoadjuvant Trastuzumab Deruxtecan (T-DXd) Monotherapy or T-DXd Followed by THP Compared to ddAC-THP in Participants With High-risk HER2-positive Early-stage Breast Cancer (DESTINY-Breast11)
Brief Title: Trastuzumab Deruxtecan (T-DXd) Alone or in Sequence With THP, Versus Standard Treatment (ddAC-THP), in HER2-positive Early Breast Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D967RC00001; 2023-505210-18-00 (Registry Identifier: CTIS (EU)); 2021-000603-21 (EudraCT Number)
Record Dates: First submitted 2021-10-22; First posted 2021-11-09 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Breast Neoplasms; Breast Cancer; HER2-positive Early Breast Cancer
Keywords: Trastuzumab Trastuzumab Deruxtecan (T-DXd; DS-8201a); DESTINY-BREAST11; Receptor, ErbB-2; breast neoplasms; Antineoplastic Agents, Phytogenic; Antineoplastic Agents;Molecular Mechanisms of Pharmacological Action; DB11; Enhertu; HER2 (human epidermal growth factor receptor 2); breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — trastuzumab deruxtecan; Paclitaxel; Trastuzumab; pertuzumab; Doxorubicin; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of three arms in parallel for the duration of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Trastuzumab deruxtecan
  Interventions: Drug: Trastuzumab Deruxtecan
- Arm B (Experimental): T-DXd, followed by THP
  Interventions: Drug: Trastuzumab Deruxtecan; Drug: Paclitaxel; Drug: Trastuzumab; Drug: Pertuzumab
- Arm C (Active Comparator): doxorubicin and cyclophosphamide, followed by THP
  Interventions: Drug: Paclitaxel; Drug: Trastuzumab; Drug: Pertuzumab; Drug: Doxorubicin; Drug: cyclophosphamide

INTERVENTIONS:
Drug: Trastuzumab Deruxtecan — administered by intravenous infusion
  Other Names: T-DXd; Enhertu
  Arms: Arm A; Arm B
Drug: Paclitaxel — administered by intravenous infusion
  Other Names: Taxol; Onxol
  Arms: Arm B; Arm C
Drug: Trastuzumab — administered by intravenous infusion
  Other Names: Herceptin; Herzuma
  Arms: Arm B; Arm C
Drug: Pertuzumab — administered by intravenous infusion
  Other Names: Perjeta
  Arms: Arm B; Arm C
Drug: Doxorubicin — administered by intravenous infusion
  Other Names: Adriamycin; Rubex
  Arms: Arm C
Drug: cyclophosphamide — administered by intravenous infusion
  Other Names: Neosar; Cytoxan
  Arms: Arm C

SUMMARY:
This study will look at the efficacy and safety of trastuzumab deruxtecan (T-DXd) in a neoadjuvant setting, in high-risk, HER2-positive early non-metastatic breast cancer.

DETAILED DESCRIPTION:
The target population of interest in this study is participants with high-risk HER2-positive early-stage breast cancer. The purpose of this study is to determine the efficacy and safety of T-DXd neoadjuvant therapy.

Participants will be randomised to one of 3 arms: T-DXd monotherapy (Arm A), T-DXd followed by THP (Arm B), or ddAC-THP (Arm C).

ELIGIBILITY:
Key Inclusion Criteria:

* Patients must be at least 18 years of age.
* Histologically documented HER2-positive early breast cancer (EBC) participants, including clinical stage at presentation (based on mammogram or breast MRI assessment): T0-4 (inclusive of inflammatory breast cancer), N1-3, M0 or ≥ T3, N0, M0 as determined by the AJCC staging system, 8th edition
* ECOG performance status of 0 or 1 at randomization
* Adequate organ and bone marrow function
* LVEF ≥ 50% within 28 days before randomization
* FFPE tissue block (2 cores) or 20 freshly-cut, serial tumor slides for HER2 assessment by central lab. If blocks are incomplete or fewer than 20 slides are available, participants may be eligible following discussion with the AstraZeneca Study Physician

Exclusion Criteria:

* prior history of invasive breast cancer
* stage IV breast cancer (determined by AJCC staging system)
* any primary malignancy within 3 years (except resected non-melanoma skin cancer, curatively treated in situ disease) Note: This includes a second current breast primary malignancy (ie, bilateral breast cancer)
* history of DCIS (except those treated with mastectomy >5 years prior to current diagnosis)
* History of, or current, ILD/pneumonitis
* Prior systemic therapy for the treatment of breast cancer
* Previous treatment with anthracyclines, cyclophosphamide or taxanes for any malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 927 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
rate of pathologic complete response (pCR) | Up to 39 months after study start
  Proportion of participants who have no evidence by H&E staining of residual invasive disease

SECONDARY OUTCOMES:
Event-Free Survival | Up to 72 months after study start
Invasive Disease-Free Survival (IDFS) | Up to 72 months after study start
Overall Survival | Up to 72 months after study start

CONTACTS AND LOCATIONS:
Locations (120):
- United States (22):
  - Research Site, Springdale, Arkansas
  - Research Site, Beverly Hills, California
  - Research Site, Glendale, California
  - Research Site, Los Alamitos, California
  - Research Site, Orange, California
  - Research Site, New Haven, Connecticut
  - Research Site, Fort Wayne, Indiana
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Shreveport, Louisiana
  - Research Site, Minneapolis, Minnesota
  - Research Site, Las Vegas, Nevada
  - Research Site, East Brunswick, New Jersey
  - Research Site, Summit, New Jersey
  - Research Site, Commack, New York
  - Research Site, Durham, North Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Germantown, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Fort Worth, Texas
  - Research Site, Ogden, Utah
  - Research Site, Tacoma, Washington
- Brazil (5):
  - Research Site, Goiânia
  - Research Site, Ijuí
  - Research Site, Natal
  - Research Site, Porto Alegre
  - Research Site, São Paulo
- Bulgaria (2):
  - Research Site, Panagyurishte
  - Research Site, Sofia
- Canada (6):
  - Research Site, Edmonton, Alberta
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Sherbrooke, Quebec
  - Research Site, Montreal
- China (12):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Kunming
  - Research Site, Nanning
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Zhengzhou
- Germany (12):
  - Research Site, Augsburg
  - Research Site, Berlin
  - Research Site, Erlangen
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Kiel
  - Research Site, Leipzig
  - Research Site, Mönchengladbach
  - Research Site, München
  - Research Site, Münster
  - Research Site, Paderborn
  - Research Site, Tübingen
- India (9):
  - Research Site, Gūrgaon
  - Research Site, Howrah
  - Research Site, Nagpur
  - Research Site, Nashik
  - Research Site, New Delhi
  - Research Site, Raipur
  - Research Site, Rishikesh
  - Research Site, Surat
  - Research Site, Thiruvananthapuram
- Italy (10):
  - Research Site, Bologna
  - Research Site, Candiolo
  - Research Site, Livorno
  - Research Site, Milan
  - Research Site, Naples
  - Research Site, Napoli
  - Research Site, Negrar
  - Research Site, Padua
  - Research Site, Roma
  - Research Site, Rozzano
- Japan (8):
  - Research Site, Chūōku
  - Research Site, Hidaka-shi
  - Research Site, Hiroshima
  - Research Site, Kawasaki-shi
  - Research Site, Kōtoku
  - Research Site, Nagoya
  - Research Site, Ota-shi
  - Research Site, Shinjuku-ku
- Research Site, Lima, Peru
- Philippines (6):
  - Research Site, Bacolod
  - Research Site, Cebu City
  - Research Site, Davao City
  - Research Site, Iloilo City
  - Research Site, Quezon City
  - Research Site, San Juan City
- Poland (7):
  - Research Site, Bialystok
  - Research Site, Biała Podlaska
  - Research Site, Bydgoszcz
  - Research Site, Koszalin
  - Research Site, Lublin
  - Research Site, Rzeszów
  - Research Site, Warsaw
- Russia (2):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Saudi Arabia (3):
  - Research Site, Dammam
  - Research Site, Jeddah
  - Research Site, Riyadh
- South Korea (2):
  - Research Site, Goyang-si
  - Research Site, Seoul
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Seville
  - Research Site, Vigo
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (4):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
  - Research Site, Hat Yai
  - Research Site, Khon Kaen

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient data from AstraZeneca Group of Companies, sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ Disclosure Commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved, AstraZeneca will provide access to the de-identified patient level data in an approved sponsor tool. Signed Data Sharing Agreements (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure